CLINICAL TRIAL: NCT03160118
Title: A Clinical Study of Biomarkers of Innate and Adaptive Immune Activation Associated with Symptoms and Immune Responses After Administration of a Single Dose of a Quadrivalent Inactivated Split Virus Influenza Vaccine to Healthy Young Adults.
Brief Title: Study of Biomarkers of Immune Activation Associated with Symptoms and Immune Responses After Influenza Vaccination in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other); Max Planck Institute for Infection Biology (MPIIB), Berlin, Germany (Unknown); deCODE genetics, Iceland (Unknown); VisMederi srl, Sienna, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BioVacSafe - QIV
Record Dates: First submitted 2017-03-24; First posted 2017-05-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Prevention of Influenza
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Seasonal,quadrivalent,influenza vaccine (Other): 1 vaccine will be administered to all participants, namely Alfa-Rix Tetra 2016-2017
  Interventions: Drug: Seasonal,quadrivalent,influenza vaccine

INTERVENTIONS:
Drug: Seasonal,quadrivalent,influenza vaccine — 1 dose to be administered on Day 0, the first visit
  Other Names: Alfa-Rix Tetra 2016-2017

SUMMARY:
This clinical fase IV study, using the administration of a single dose of a quadrivalent, inactivated, split influenza virus vaccine as biological intervention will mirror a study conducted at Imperial College, London, UK that will use a challenge with live virus as intervention. Comparison of the clinical observations and laboratory measurements generated in both studies will inform us about the similarities and differences in innate and adaptive immune responses elicited by both types of exposure to influenza virus antigen(s).

DETAILED DESCRIPTION:
The study is a monocentric, open label study. All subjects will receive a single dose of alfa-Rix Tetra 2016-2017. The following will be measured - clinical events (recorded adverse events), physiological responses (heart rate, blood pressure, temperature, injection site), innate immune responses (cytokine levels and whole blood gene expression) and adaptive immune responses (serum antibody and antigen-specific cellular responses) at various time points after immunisation.

At each study visit, full physiological parameters (including body temperature, heart rate, blood pressure) will be obtained and the injection site will be examined for the presence of any redness or swelling that will be measured and recorded. Standardized diary cards will be used to collect solicited and unsolicited clinical event data. At each visit the diary cards will be examined and any relevant clinical event will be entered into the clinical event form. Participants will be asked to monitor oral temperature from day 0 until day 7 when they wake up and when going to bed. The results of these measurements will be reported in a diary card. Any skin reactions at the site of injection will be evaluated; largest diameter of redness and swelling will be measured with a ruler and data reported on the diary card. Samples of blood (PAXgene tubes, plasma, serum and PBMCs (peripheral blood mononuclear cells)) will be collected for analysis and processing using protocols already in place. Subjects will also have blood obtained for standard safety markers (haematology, biochemistry) as well as acute phase proteins.

The purpose of this protocol is to generate a set of data that will be analysed by integrated systems biology approach, for validation in subsequent clinical trials or in animal models. The dataset will broadly characterise:

1. Physiological responses at various time points after immunisation by measuring:

   1. Local and systemic vaccine-related clinical events.
   2. Physiological assessments: heart rate, body temperature, blood pressure.
   3. Haematology (Complete Blood Count (CBC), Erythrocyte Sedimentation Rate (ESR) , phenotyping of White Blood Cells (WBC)), biochemistry parameters.
2. Innate and adaptive immune responses including:

   1. Innate immune activation detected by global gene expression in whole blood
   2. Adaptive immunity determined by:

   i. Humoral immune response via serum anti-influenza HAI (Haemagglutination Inhibition) titre ii. Cellular immune response c. Immune activation detected by concentration of selected inflammatory soluble mediators in serum including: i. chemokines and cytokines ii. acute phase proteins
3. Genetic testing of subjects when deemed necessary (genetic testing analysis may be SNIP (Single Nucleotide Polymorphism) analysis or full genome analysis).
4. Correlations in changes in innate and adaptive immune activation with adverse events, haematology and biochemistry panels, genotype and physiological assessments

The study team will biobank all samples for the duration of the BIOVACSAFE programme so that different samples and different time points depending on the results generated can selectively be analysed, principally from the gene expression analysis of whole blood.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged 24-54 years inclusive. (Healthy in the opinion of the investigator, based on medical history and clinical exam, with no active disease process that could interfere with the study endpoints)
2. Has a body Mass Index ≥18 and ≤30
3. Is able to read and understand the Informed Consent Form (ICF), and understand study procedures.
4. The subject has signed the ICF.
5. The subject is available for follow-up for the duration of the study.
6. The subject agrees to abstain from donating blood during their participation in the study, or longer if necessary.
7. If the subject is a heterosexually active female, she is willing to use an effective method of contraception (e.g. oral contraceptive pill; intrauterine device; injectable or implanted contraceptive; physiological or anatomical sterility) from 30 days prior to study vaccination until the end of the study.
8. Willing to undergo urine pregnancy tests prior to vaccination at screening.
9. The subject has venous access sufficient to allow blood sampling as per the protocol.

Exclusion Criteria:

1. Pregnant or lactating.
2. Known hypersensitivity to any component of the study vaccine (α-RIX-Tetra®): the active components (vaccine antigens) or any of the excipients (disodium phosphate dodecahydrate, potassium dihydrogen phosphate, magnesium chloride hexahydrate, α-tocopheryl hydrogen succinate, polysorbate 80, octoxinol 10), eggs (chicken proteins, ovalbumin), gentamycin sulphate, formaldehyde, and sodium deoxycholate or those who have had a previous life-threatening reaction to previous influenza vaccinations.
3. History of influenza infection in the past 5 years, defined here as severe respiratory infection with fever (> 38°C) and preventing normal daily activity during a minimum of 3 days.
4. Vaccination with the 2016/2017 seasonal influenza vaccine and/or any other seasonal influenza vaccine within the preceding 5 influenza seasons (i.e. since season 2011/2012) before the first study visit.
5. Presence of primary or acquired immunodeficiency states with a total lymphocyte count less than 1,200 per mm3 or presenting other evidence of lack of cellular immune competence e.g. leukaemias, lymphomas, blood dyscrasias, or patients receiving immunosuppressive therapy (including use of oral or parenteral corticosteroids in a dose ≥ 5 mg prednisone daily or equivalent within one month prior to visit 1or cytotoxic or immunosuppressive or immunomodulating drugs within 6 months prior to visit 1).
6. Regular use of non-steroidal anti-inflammatory drugs (oral or parenteral route) within 6 months of Visit 1 considered by the study physician as likely to interfere with immune responses.
7. Current intake of excessive amounts of alcohol (≥ 14 units for women and ≥ 21 units for men) and not willing to adapt this use during the study period.
8. Currently performing extreme physical activities (as evaluated by the investigator) and not willing to adapt this activity during the study period.
9. Receipt of a vaccine within 30 days of visit 1, or requirement to receive another vaccine within the study period.
10. Presence of an acute severe febrile illness at time of immunisation.
11. History of alcohol, narcotic, benzodiazepine, rilatine, or other substance abuse or dependence within the 12 months preceding Visit 1.
12. Smoking in the past 6 months OR > 5 pack-year lifetime history
13. Receipt of blood products or immunoglobulins, or blood donation, within 3 months of study start.
14. Any condition that, in the investigator's opinion, compromises the subject's ability to meet protocol requirements or to complete the study.
15. Currently participating in another clinical study with an investigational or non-investigational drug or device, or has participated in a clinical trial within the 3 months preceding Visit 1.
16. Unable to read and speak Dutch or English to a fluency level adequate for the full comprehension of procedures required in participation and consent.

Ages: 24 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-06-28 (Actual)

PRIMARY OUTCOMES:
Frequency of local vaccine-related clinical events. | At all timepoints from vaccination up to 28 days after vaccination
  Participants will report these events on a diary, measuring local events or scoring them from 0 (absent) to 3 (severe)
Severity of local vaccine-related clinical events. | At all timepoints from time of vaccination up to 28 days after vaccination
  Participants will report these events on a diary, measuring local events or scoring them from 0 (absent) to 3 (severe)
Frequency of systemic vaccine-related clinical events. | At selected timepoints from time of vaccination up to 28 days after vaccination
  Participants will report these events on a diary, scoring the events from 0 (absent) to 3 (severe)
Severity of systemic vaccine-related clinical events. | At selected timepoints from time of vaccination up to 28 days after vaccination
  Participants will report these events on a diary, scoring the events from 0 (absent) to 3 (severe)
Change from pre-immunisation baseline values in pulse. | At selected timepoints from time of vaccination up to 28 days after vaccination
  Will be measured during the study visits
Change from pre-immunisation baseline values in body temperature | At selected timepoints from time of vaccination up to 28 days after vaccination
  Will be measured during the study visits
Change from pre-immunisation baseline values in blood pressure | At selected timepoints from time of vaccination up to 28 days after vaccination
  Will be measured during the study visits
Change from pre-immunisation baseline values in haematology (CBC, ESR, phenotyping of WBC) parameters | At selected timepoints from time of vaccination up to 28 days after vaccination
  blood will be collected during the study visits
Change from pre-immunisation baseline values in biochemistry parameters | At selected timepoints from time of vaccination up to 28 days after vaccination
  blood will be collected during the study visits
Change from pre-immunisation baseline values in global gene expression measured on whole blood samples | At selected timepoints from time of vaccination up to 28 days after vaccination
  blood will be collected during the study visits
Change from pre-immunisation baseline values in serum HAI titre in serum samples | At selected timepoints from time of vaccination up to 28 days after vaccination
  blood will be collected during the study visits
Change from pre-immunisation values of adaptive cellular immune response via enumeration of influenza-specific CD4+ T cells expressing activation markers and/or cytokines following in vitro stimulation and analysis by flow cytometry | At selected timepoints from time of vaccination up to 28 days after vaccination
  blood will be collected during the study visits
Change from pre-immunisation baseline values in concentration of selected cytokines and acute phase proteins in serum samples | At selected timepoints from time of vaccination up to 28 days after vaccination
  blood will be collected during the study visits
Change from pre-immunisation baseline values in PBMC cytokine secretion, proliferation or surface markers in response to in vitro stimulation with influenza antigens | At selected timepoints from time of vaccination up to 28 days after vaccination
  blood will be collected during the study visits

CONTACTS AND LOCATIONS:
Overall Officials: Geert Leroux-Roels, Prof., PhD, Principal Investigator — University Ghent / University Hospital Ghent
Locations (1):
- University Hospital - Center for Vaccinology, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No